CLINICAL TRIAL: NCT00280059
Title: A Randomized, Comparative, Double-Blind, Parallel-Group, Multicenter, Monotherapy, Study Of Pregabalin (Lyrica) And Lamotrigine (Lamictal) In Patients With Newly Diagnosed Partial Seizures
Brief Title: Study Of The Safety And Efficacy Of Lyrica In The Treatment Of Newly Diagnosed Partial Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0081046
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Results first posted 2011-10-24 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2015-03

CONDITIONS: Epilepsy, Partial
Keywords: Epilepsy; partial seizures; pregabalin monotherapy; lamotrigine comparator; double-blind and randomized trial
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Seizures | interventions — Pregabalin; Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Pregabalin
- 2 (Active Comparator)
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Pregabalin — dose 150-600 mg/day given BID
  Arms: 1
Drug: Lamotrigine — dose 100-500 mg/day given BID
  Arms: 2

SUMMARY:
The purpose of this study is to assess whether Lyrica is a safe and effective treatment for partial epilepsy in comparison with an established treatment, Lamictal.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with partial epilepsy and have experienced at least 2 partial seizures (simple partial, complex partial or partial seizure with secondary generalization) in the past year with one in the past 6 months.

Exclusion Criteria:

* Treatable causes of seizures, for example identified etiologies including metabolic, neoplastic or active infectious origin.
* Primary generalized seizures.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2006-08; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (85):
- Belgium (3):
  - Pfizer Investigational Site, Bruges
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Leuven
- Bulgaria (3):
  - Pfizer Investigational Site, Plovdiv
  - Pfizer Investigational Site, Sofia
  - Pfizer Investigational Site, Varna
- China (4):
  - Pfizer Investigational Site, Xi’an, Shanxi
  - Pfizer Investigational Site, Cheng Du Si Chaun
  - Pfizer Investigational Site, Chongqing
  - Pfizer Investigational Site, Tianjin
- Colombia (2):
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Cali, Valle del Cauca Department
- Czechia (7):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Ostrava
  - Pfizer Investigational Site, Pelhřimov
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Rychnov nad Kněžnou
  - Pfizer Investigational Site, Zlín
- Estonia (2):
  - Pfizer Investigational Site, Tallinn
  - Pfizer Investigational Site, Tartu
- Finland (2):
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Tampere
- France (3):
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Nancy
  - Pfizer Investigational Site, Strasbourg
- Germany (5):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Ulm
- Hong Kong (3):
  - Pfizer Investigational Site, Hong Kong
  - Pfizer Investigational Site, Kowloon
  - Pfizer Investigational Site, Shatin
- Hungary (3):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Győr
  - Pfizer Investigational Site, Nyíregyháza
- India (6):
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Indore, Madhya Pradesh
  - Pfizer Investigational Site, Chennai, Tamil Nadu
  - Pfizer Investigational Site, Bangalore
  - Pfizer Investigational Site, Lucknow
  - Pfizer Investigational Site, New Delhi
- Pfizer Investigational Site, Tallaght, Dublin, Ireland
- Italy (4):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Foggia
  - Pfizer Investigational Site, Pisa
- Pfizer Investigational Site, Riga, Latvia
- Lithuania (2):
  - Pfizer Investigational Site, Kaunas
  - Pfizer Investigational Site, Vilnius
- Mexico (2):
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, San Luis Potosí City
- Pfizer Investigational Site, The Hague, South Holland, Netherlands
- Norway (2):
  - Pfizer Investigational Site, Lillehammer
  - Pfizer Investigational Site, Trondheim
- Portugal (3):
  - Pfizer Investigational Site, Amadora
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Porto
- Romania (2):
  - Pfizer Investigational Site, Cluj-Napoca, Jud. Cluj
  - Pfizer Investigational Site, Bucharest
- Pfizer Investigational Site, Singapore, Singapore
- Slovakia (3):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Košice
  - Pfizer Investigational Site, Žilina
- South Korea (4):
  - Pfizer Investigational Site, Daejeon
  - Pfizer Investigational Site, Gwangju
  - Pfizer Investigational Site, Incheon
  - Pfizer Investigational Site, Seoul
- Spain (4):
  - Pfizer Investigational Site, Badalona, Barcelona
  - Pfizer Investigational Site, Girona
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Valencia
- Sweden (3):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Uppsala
- Taiwan (2):
  - Pfizer Investigational Site, Tainan
  - Pfizer Investigational Site, Taipei
- Thailand (3):
  - Pfizer Investigational Site, Rajthevee, Bangkok
  - Pfizer Investigational Site, Muang, Changwat Khon Kaen
  - Pfizer Investigational Site, Bangkok
- United Kingdom (4):
  - Pfizer Investigational Site, Stoke-on-Trent, Staffordshire
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Liverpool
  - Pfizer Investigational Site, Treliske, Truro, Cornwall

REFERENCES:
- [Derived] Kwan P, Brodie MJ, Kalviainen R, Yurkewicz L, Weaver J, Knapp LE. Efficacy and safety of pregabalin versus lamotrigine in patients with newly diagnosed partial seizures: a phase 3, double-blind, randomised, parallel-group trial. Lancet Neurol. 2011 Oct;10(10):881-90. doi: 10.1016/S1474-4422(11)70154-5. Epub 2011 Aug 31. PMID 21889410
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081046&StudyName=Study%20Of%20The%20Safety%20And%20Efficacy%20Of%20Lyrica%20In%20The%20Treatment%20Of%20Newly%20Diagnosed%20Partial%20Epilepsy

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin: Pregabalin 150, 300, 450 or 600 mg/day orally twice daily (BID); individual titration based on number of seizures experienced once Level 1 (150 mg/day) was maintained for at least 7 days, and dose reductions based on intolerable adverse events. Escalation to next dose level allowed only after completing previous dose level for at least 1 week.
- Lamotrigine: Lamotrigine 100, 200, 400, or 500 mg/day orally BID; individual titration based on number of seizures experienced once Level 1 (100 mg/day) was reached and maintained for 7 days, and dose reductions based on intolerable adverse events. Escalation to next dose level allowed only after completing previous dose level for at least 1 week.
Period: Efficacy Assessment Phase
Arm/Group | Pregabalin | Lamotrigine
Started | 330 | 330
Completed | 236 (Week 56: up to end of efficacy assessment phase (excluding extension phase).) | 250 (Week 56: up to end of efficacy assessment phase (excluding extension phase).)
Not Completed | 94 | 80
Not completed — Death | 2 | 0
Not completed — Adverse Event | 33 | 31
Not completed — Laboratory abnormaility | 1 | 0
Not completed — Lack of Efficacy | 19 | 3
Not completed — Lost to Follow-up | 6 | 13
Not completed — Other | 7 | 8
Not completed — Withdrawal by Subject | 26 | 25
Period: Extension Phase
Arm/Group | Pregabalin | Lamotrigine
Started | 194 (Optional phase; number entered was less than the number who completed the efficacy assessment phase.) | 215 (Optional phase; number entered was less than the number who completed the efficacy assessment phase.)
Completed | 145 | 177
Not Completed | 49 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Lamotrigine | Total
Number analyzed (Participants) | 330 | 330 | 660
Age, Customized [Number; unit: participants]
  < 18 years | 9 | 9 | 18
  Between 18 and 44 years | 228 | 228 | 456
  Between 45 and 64 years | 79 | 74 | 153
  >= 65 years | 14 | 19 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 146 | 311
  Male | 165 | 184 | 349

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Seizure-free Participants (Responders) During Efficacy Assessment Phase
Description: Responders = participants who achieved any 6 consecutive months (>182 days) of seizure-freedom (absence of partial seizures, generalized seizures and unclassified epileptic seizures) during the 52 week efficacy assessment phase.
Time Frame: Week 5 up to Week 56
Population: Full analysis set (FAS) (intent to treat population): randomized participants who took at least 1 dose of study medication. N = number of participants who had at least 1 dose of study treatment and seizure efficacy data. Analysis excludes participants who did not enter maintenance phase of study.
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 314 | 308
percentage of participants | 51.6 | 67.9
Statistical Analysis 1: Comparison: Pregabalin vs Lamotrigine; Analysis of the binary response variable for 6 consecutive months seizure freedom analyzed by comparing the proportions of favorable responders between the two treatment groups after stratifying by clusters and correcting for skewness (Gart and Nam, 1990). Percentage can be obtained by multiplying proportion by 100; Test type: Non-Inferiority or Equivalence — Non-inferiority margin for the proportion of seizure free participants set at 10%; non-inferiority declared if the lower bound of the 95% confidence interval (CI) of the difference in seizure-free proportion between pregabalin and lamotrigine was no more than 10% in favor of lamotrigine, but 0 was contained within the lower bound of the CI. Interpretation of superiority required lower bound of CI did not contain 0 in favor of pregabalin; Gart and Nam: correction of skewness; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.24 to -0.09] — 95% confidence interval for the true difference in proportions, as well as a one-sided test at α=0.025; confidence interval adjusted for centers clustered within a geographical region, with upper and lower confidence limits

2. Secondary Outcome: Time to 6 Consecutive Months of Seizure-freedom After 4-week Dose Escalation Phase: All Seizures
Description: Time in days, from first day of study medication to the first 6 months of seizure freedom after Day 28. Participants who did not achieve 6 months seizure freedom after Day 28 were censored from analysis.
Time Frame: Week 4 up to Week 56
Population: FAS. N = number of participants who entered maintenance phase of study and had seizure efficacy data.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 314 | 308
days | 254 [199 to 295] | 183 [183 to 209]
Statistical Analysis 1: Comparison: Pregabalin vs Lamotrigine; Risk ratio=hazard ratio estimated from the Cox proportional hazards model for assessing a treatment difference, risk ratio > 1 is in favor of pregabalin. The 95% confidence interval is for the true risk ratio; Test type: Superiority or Other; p = 0.0034, Regression, Cox — Nominal value for 2-sided test calculated using Cox proportional hazards model, adjusted for geographic regions; Risk Ratio (RR) = 0.74, 95% CI 2-sided [0.60 to 0.90]

3. Secondary Outcome: Exit Due to Adverse Events During the Double-blind Treatment Phase (Including Dose Escalation Phase)
Description: Number of participants who exited the study due to adverse events during the double-blind treatment period. Time in days, from first day of study treatment to day of exit from the study due to an adverse event (ie, last day on study medication) during the double blind treatment period (including dose escalation phase) was inestimable. Observations with other reasons for exiting or participants who did not exit the study were right censored as of the last day on study medication.
Time Frame: Week 0 to Week 56
Population: FAS. N = number of participants who entered maintenance phase of study and had seizure efficacy data. Time to exit due to adverse events was inestimable as survival estimate at end of maintenance phase was below 0.500.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 330 | 330
participants | 33 | 31
Statistical Analysis 1: Comparison: Pregabalin vs Lamotrigine; Risk ratio=hazard ratio estimated from the Cox proportional hazards model for assessing a treatment difference, risk ratio < 1 is in favor of pregabalin. The 95% confidence interval is for the true risk ratio; Test type: Superiority or Other; p = 0.8047, Cox proportional hazards model — Nominal value for 2-sided test calculated using Cox proportional hazards model adjusted for geographical cluster; Risk Ratio (RR) = 1.06, 95% CI 2-sided [0.65 to 1.74]

4. Secondary Outcome: Exit for Any Reason During the Double-blind Treatment Phase (Including Dose Escalation Phase)
Description: Number of participants who exited the study for any reason during the double blind treatment phase. Time in days, from first day of study treatment to day of exit from the study due to any reason (ie, last day on study medication) was inestimable. Participants who did not exit the study were right censored as of the last day on study medication.
Time Frame: Week 0 to Week 56
Population: FAS. N = number of participants who had at least 1 dose of study treatment and seizure efficacy data Time to exit for any reason during the double-blind treatment phase was inestimable as the survival estimate at the end of the maintenance phase was below 0.500.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 330 | 330
participants | 94 | 80
Statistical Analysis 1: Comparison: Pregabalin vs Lamotrigine; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2537, Cox proportional hazards model — Nominal value for 2-sided test calculated using Cox proportional hazards model adjusted for geographical cluster; Risk Ratio (RR) = 1.19, 95% CI 2-sided [0.88 to 1.60]

5. Secondary Outcome: Exit Due to Lack of Efficacy After 4-week Dose Escalation Phase
Description: Number of participants who exited the study due to lack of efficacy after the 4-week dose escalation phase. Time in days, from first day of study treatment to day of exit due to lack of efficacy after Day 28 of the escalation phase (ie, last day on study medication) was inestimable. Participants who did not exit or exited for a different reason were right censored as of the last day on study medication.
Time Frame: Week 4 up to Week 56
Population: FAS. N = number of participants who entered maintenance phase of study and had seizure efficacy data. Time to exit due to lack of efficacy after 4-week dose escalation phase was inestimable as survival estimate at end of maintenance phase was below 0.500.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 329 | 330
participants | 78 | 58
Statistical Analysis 1: Comparison: Pregabalin vs Lamotrigine; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0025, Cox proportional hazards model — Nominal value for 2-sided test calculated using Cox proportional hazards model adjusted for geographical cluster; Risk Ratio (RR) = 6.52, 95% CI 2-sided [1.93 to 22.04]

6. Secondary Outcome: Exit Due to Any Reason After 4-week Dose Escalation Phase
Description: Number of participants who exited the study due to any reason after the 4-week dose escalation phase. Time in days, from first day of study treatment to day of exit after Day 28 of the study due to any reason (ie, last day on study medication) was inestimable. Participants who did not exit or did not reach this phase were right censored as of the last day on study medication.
Time Frame: Week 4 up to Week 56
Population: FAS. N = number of participants who entered maintenance phase of study and had seizure efficacy data. Time to exit for any reason after the 4-week dose escalation phase was inestimable as the survival estimate at the end of the maintenance phase was below 0.500.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 329 | 300
participants | 78 | 58
Statistical Analysis 1: Comparison: Pregabalin vs Lamotrigine; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0744, Cox proportional hazards model — Nominal value for 2-sided test calculated using Cox proportional hazards model adjusted for geographical cluster; Risk Ratio (RR) = 1.36, 95% CI 2-sided [0.97 to 1.91]

7. Secondary Outcome: Time to First Seizure After the 4-Week Dose Escalation Phase
Description: Time in days, from first day of study treatment to the day of first seizure after Day 28 of the escalation phase (ie, last day on study medication). Participants who did not reach this phase or who did not have a seizure after Day 28 were right censored from the analysis as of the last day on study medication.
Time Frame: Week 4 up to Week 56
Population: FAS. N = number of participants who entered maintenance phase of study and had seizure efficacy data.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 329 | 300
days | 85 [59 to 120] | 211 [145 to 342]
Statistical Analysis 1: Comparison: Pregabalin vs Lamotrigine; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0003, Cox proportional hazards model — Nominal value for 2-sided test calculated using Cox proportional hazards model adjusted for geographical cluster; Risk Ratio (RR) = 1.47, 95% CI 2-sided [1.19 to 1.80]

8. Secondary Outcome: Median Monthy Seizure Frequency: All Partial Seizures
Description: All partial seizures include complex partial seizures, simple partial seizures, and partial seizures evolving to secondarily generalized seizures. Seizure frequency based on 28-day seizure rate: number (#) of seizures in period (month) divided by # days in period minus # of missing diary days in period * 28. Month of time = number of months after Week 4 (Dose Escalation).
Time Frame: Baseline up to Week 60
Population: FAS. N = number of participants with analyzable data; n = number of participants with analyzable data at observation.
Measure: Median (Standard Deviation); unit: seizures/28 days
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 329 | 330
seizures/28 days
  Dose-escalation phase (Weeks 1 - 4) (n=329, 330) | 0.0 (9.348) | 0.0 (27.118)
  Month 1 (n=314, 308) | 0.0 (6.139) | 0.0 (31.453)
  Month 2 (n=300, 295) | 0.0 (3.382) | 0.0 (28.839)
  Month 3 (n=287, 288) | 0.0 (2.568) | 0.0 (32.783)
  Month 4 (n=279, 278) | 0.0 (2.313) | 0.0 (16.046)
  Month 5 (n=274, 276) | 0.0 (2.270) | 0.0 (15.254)
  Month 6 (n=266, 272) | 0.0 (2.702) | 0.0 (15.126)
  Month 7 (n=260, 270) | 0.0 (2.839) | 0.0 (16.855)
  Month 8 (n=256, 266) | 0.0 (3.247) | 0.0 (19.111)
  Month 9 (n=253, 262) | 0.0 (2.538) | 0.0 (17.204)
  Month 10 (n=250, 257) | 0.0 (4.935) | 0.0 (16.905)
  Month 11 (n=242, 254) | 0.0 (3.082) | 0.0 (19.268)
  Month 12 (n=238, 252) | 0.0 (7.018) | 0.0 (19.590)
  Month 13 (n=210, 227) | 0.0 (3.247) | 0.0 (19.462)
  Taper (Week 57 to Week 60) (n=71, 45) | 0.0 (6.418) | 0.0 (97.196)

9. Secondary Outcome: Mean Monthy Seizure Frequency: All Partial Seizures
Description: as for outcome 8
Time Frame: Baseline up to Week 60
Population: FAS. N = number of participants with analyzable data; n = number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: seizures/28 days
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 329 | 330
seizures/28 days
  Dose escalation phase (n=329, 330) | 2.56 (9.348) | 5.08 (27.118)
  Month 1 (n=314, 308) | 2.23 (6.139) | 4.21 (31.453)
  Month 2 (n=300, 295) | 1.18 (3.382) | 3.21 (28.839)
  Month 3 (n=287, 288) | 0.94 (2.568) | 3.54 (32.783)
  Month 4 (n=279, 278) | 0.89 (2.313) | 1.67 (16.046)
  Month 5 (n=274, 276) | 0.78 (2.270) | 1.58 (15.254)
  Month 6 (n=266, 272) | 0.82 (2.702) | 1.41 (15.126)
  Month 7 (n=260, 270) | 0.78 (2.839) | 1.50 (16.855)
  Month 8 (n=256, 266) | 0.77 (3.247) | 1.36 (19.111)
  Month 9 (n=253, 262) | 0.71 (2.538) | 1.38 (17.204)
  Month 10 (n=250, 257) | 1.05 (4.935) | 1.33 (16.905)
  Month 11 (n=242, 254) | 0.79 (3.082) | 1.41 (19.268)
  Month 12 (n=238, 252) | 0.94 (7.018) | 1.67 (19.590)
  Month 13 (n=210, 227) | 0.65 (3.247) | 2.11 (19.462)
  Taper (n=71, 45) | 2.13 (6.418) | 19.97 (97.196)

10. Secondary Outcome: Median Monthy Seizure Frequency: All Seizures
Description: Seizure frequency based on 28-day seizure rate: number (#) of seizures in period (month) divided by # days in period minus # of missing diary days in period * 28. Month of time = number of months after Week 4 (Dose Escalation).
Time Frame: Baseline up to Week 60
Population: FAS. N = number of participants with analyzable data; n = number of participants with analyzable data at observation.
Measure: Median (Standard Deviation); unit: seizures/28 days
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 329 | 330
seizures/28 days
  Dose-escalation phase (Weeks 1 - 4)(n=329, 330) | 0.0 (9.819) | 0.0 (27.128)
  Month 1 (n=314, 308) | 0.0 (6.164) | 0.0 (31.452)
  Month 2 (n=300, 295) | 0.0 (5.498) | 0.0 (28.838)
  Month 3 (n=287, 288) | 0.0 (2.702) | 0.0 (32.782)
  Month 4 (n=279, 278) | 0.0 (3.223) | 0.0 (16.046)
  Month 5 (n=274, 276) | 0.0 (2.458) | 0.0 (15.254)
  Month 6 (n=266, 272) | 0.0 (2.853) | 0.0 (15.126)
  Month 7 (n=260, 270) | 0.0 (2.898) | 0.0 (16.855)
  Month 8 (n=256, 266) | 0.0 (3.304) | 0.0 (19.110)
  Month 9 (n=253, 262) | 0.0 (2.636) | 0.0 (17.204)
  Month 10 (n=250, 257) | 0.0 (4.934) | 0.0 (16.905)
  Month 11 (n=242, 254) | 0.0 (3.224) | 0.0 (19.268)
  Month 12 (n=238, 252) | 0.0 (7.019) | 0.0 (19.590)
  Month 13 (n=210, 227) | 0.0 (3.247) | 0.0 (19.462)
  Taper (Week 57 to Week 60) (n=71, 45) | 0.0 (6.418) | 0.0 (97.196)

11. Secondary Outcome: Mean Monthy Seizure Frequency: All Seizures
Description: as for outcome 10
Time Frame: Baseline up to Week 60
Population: FAS. N = number of participants with analyzable data; n = number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: seizures/28 days
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 329 | 330
seizures/28 days
  Dose-escalation phase (n=329, 330) | 2.74 (9.819) | 5.10 (27.128)
  Month 1 (n=314, 308) | 2.31 (6.164) | 4.24 (31.452)
  Month 2 (n=300, 295) | 1.53 (5.498) | 3.22 (28.838)
  Month 3 (n=287, 288) | 1.02 (2.702) | 3.57 (32.782)
  Month 4 (n=279, 278) | 1.06 (3.223) | 1.68 (16.046)
  Month 5 (n=274, 276) | 0.87 (2.458) | 1.59 (15.254)
  Month 6 (n=266, 272) | 0.89 (2.853) | 1.41 (15.126)
  Month 7 (n=260, 270) | 0.83 (2.898) | 1.50 (16.855)
  Month 8 (n=256, 266) | 0.82 (3.304) | 1.37 (19.110)
  Month 9 (n=253, 262) | 0.78 (2.636) | 1.38 (17.204)
  Month 10 (n=250, 257) | 1.06 (4.934) | 1.33 (16.905)
  Month 11 (n=242, 254) | 0.81 (3.224) | 1.41 (19.268)
  Month 12 (n=238, 252) | 0.96 (7.019) | 1.67 (19.590)
  Month 13 (n=210, 227) | 0.65 (3.247) | 2.12 (19.462)
  Taper (n=71, 45) | 2.13 (6.418) | 19.97 (97.196)

12. Secondary Outcome: Median Monthy Seizure Frequency of Responders for the Months After Achieving 6 Consecutive Months of Seizure Freedom: All Partial Seizures
Description: All partial seizures include complex partial seizures, simple partial seizures, and partial seizures evolving to secondarily generalized seizures. Seizure frequency based on 28-day seizure rate: number (#) of seizures in period (month) divided by # days in period minus # of missing diary days in period * 28. Responder = participant who achieved at least 6 months of seizure freedom after Week 4 and up to Week 56. Monthly seizure frequency measured from day of achievement of 6 months of seizure freedom.
Time Frame: Month 1 through Month 9 (after 6 months seizure freedom achieved)
Population: FAS. N = number of responders; n = number of responders with analyzable data at observation.
Measure: Median (Standard Deviation); unit: seizures/28 days
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 162 | 208
seizures/28 days
  Month 1 (n=162, 208) | 0.0 (1.000) | 0.0 (0.226)
  Month 2 (n=155, 194) | 0.0 (1.783) | 0.0 (0.226)
  Month 3 (n=147, 184) | 0.0 (0.384) | 0.0 (0.439)
  Month 4 (n=139, 173) | 0.0 (0.329) | 0.0 (0.211)
  Month 5 (n=127, 158) | 0.0 (0.926) | 0.0 (0.823)
  Month 6 (n=122, 152) | 0.0 (0.156) | 0.0 (0.213)
  Month 7 (n=105, 136) | 0.0 (0.000) | 0.0 (2.843)
  Month 8 (n=1, 5) | 0.0 (NA) — n = 1. | 0.0 (0.000)
  Month 9 (n=0, 1) | NA (NA) — No responders with analyzable data at Month 9. | 6.0 (NA) — n = 1.

13. Secondary Outcome: Mean Monthy Seizure Frequency of Responders for the Months After Achieving 6 Consecutive Months of Seizure Freedom: All Partial Seizures
Description: as for outcome 12
Time Frame: Month 1 through Month 9 (after 6 months seizure freedom achieved)
Population: FAS. N = number of responders; n = number of responders with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: 28-day seizure rate
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 162 | 208
28-day seizure rate
  Month 1 (n=162, 208) | 0.19 (1.000) | 0.04 (0.226)
  Month 2 (n=155, 194) | 0.28 (1.783) | 0.03 (0.226)
  Month 3 (n=147, 184) | 0.05 (0.384) | 0.07 (0.439)
  Month 4 (n=139, 173) | 0.09 (0.329) | 0.05 (0.211)
  Month 5 (n=127, 158) | 0.15 (0.926) | 0.10 (0.823)
  Month 6 (n=122, 152) | 0.02 (0.156) | 0.03 (0.213)
  Month 7 (n=105, 136) | 0.00 (0.000) | 0.28 (2.843)
  Month 8 (n=1, 5) | 0.00 (NA) — Measure of dispersion cannot be calculated with a sample size of 1. | 0.00 (0.000)
  Month 9 (n=0, 1) | NA (NA) — No responders with analyzable data at Month 9. | 6.00 (NA) — Measure of dispersion cannot be calculated with a sample size of 1.

14. Secondary Outcome: Median Monthy Seizure Frequency of Responders for the Months After Achieving 6 Consecutive Months of Seizure Freedom: All Seizures
Description: Seizure frequency based on 28-day seizure rate: number (#) of seizures in period (month) divided by # days in period minus # of missing diary days in period * 28. Responder = participant who achieved at least 6 months of seizure freedom after Week 4 and up to Week 56. Monthly seizure frequency measured from day of achievement of 6 months of seizure freedom.
Time Frame: Month 1 through Month 9 (after 6 months seizure freedom achieved)
Population: FAS. N = number of responders; n = number of responders with analyzable data at observation.
Measure: Median (Standard Deviation); unit: seizures/28 days
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 162 | 208
seizures/28 days
  Month 1 (n=162, 208) | 0.0 (1.000) | 0.0 (0.236)
  Month 2 (n=155, 194) | 0.0 (1.783) | 0.0 (0.226)
  Month 3 (n=147, 184) | 0.0 (0.400) | 0.0 (0.439)
  Month 4 (n=139, 173) | 0.0 (0.359) | 0.0 (0.211)
  Month 5 (n=127, 158) | 0.0 (0.971) | 0.0 (0.823)
  Month 6 (n=122, 152) | 0.0 (0.156) | 0.0 (0.213)
  Month 7 (n=105, 136) | 0.0 (0.000) | 0.0 (2.844)
  Month 8 (n=1, 5) | 0.0 (NA) — n=1. | 0.0 (0.000)
  Month 9 (n=0, 1) | NA (NA) — No responders with analyzable data at Month 9. | 6.0 (NA) — n=1.

15. Secondary Outcome: Mean Monthy Seizure Frequency of Responders for the Months After Achieving 6 Consecutive Months of Seizure Freedom: All Seizures
Description: as for outcome 14
Time Frame: Month 1 through Month 9 (after 6 months seizure freedom achieved)
Population: FAS. N = number of responders; n = number of responders with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: 28-day seizure rate
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 162 | 208
28-day seizure rate
  Month 1 (n=162, 208) | 0.19 (1.000) | 0.05 (0.236)
  Month 2 (n=155, 194) | 0.28 (1.783) | 0.03 (0.226)
  Month 3 (n=147, 184) | 0.07 (0.400) | 0.07 (0.439)
  Month 4 (n=139, 173) | 0.09 (0.359) | 0.05 (0.211)
  Month 5 (n=127, 158) | 0.18 (0.971) | 0.10 (0.823)
  Month 6 (n=122, 152) | 0.02 (0.156) | 0.03 (0.213)
  Month 7 (n=105, 136) | 0.00 (0.000) | 0.29 (2.844)
  Month 8 (n=1, 5) | 0.00 (NA) — Measure of dispersion cannot be calculated with a sample size of 1. | 0.00 (0.000)
  Month 9 (n=0, 1) | NA (NA) — No responders with analyzable data at Month 9. | 6.00 (NA) — Measure of dispersion cannot be calculated with a sample size of 1.

16. Secondary Outcome: Percentage of Participants Who Achieved at Least 6 Consecutive Months of Seizure Freedom (Responders) by Final Dosage Levels and Treatment Group
Description: Responder = participant who achieved at least 6-months of seizure freedom (all seizures) after Week 4, and up to Week 56. Dose Level defined as last total-daily-dose received after Week 4, and up to Week 56.
Time Frame: Week 5 up to Week 56
Population: FAS; N = number of participants with analyzable data.
Measure: Number; unit: percentage of participants
Groups:
- Pregabalin 150 mg/Day: Pregabalin 150 mg/day administered twice daily (BID)
- Pregabalin 300 mg/Day: Pregabalin 300 mg/day administered BID
- Pregabalin 450 mg/Day: Pregabalin 450 mg/day administered BID
- Pregabalin 600 mg/Day: Pregabalin 600 mg/day administered BID
- Lamotrigine 100 mg/Day: Lamotrigine 100 mg/day administered BID
- Lamotrigine 200 mg/Day: Lamotrigine 200 mg/day administered BID
- Lamotrigine 400 mg/Day: Lamotrigine 400 mg/day administered BID
- Lamotrigine 500 mg/Day: Lamotrigine 500 mg/day administered BID
Arm/Group | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregabalin 450 mg/Day | Pregabalin 600 mg/Day | Lamotrigine 100 mg/Day | Lamotrigine 200 mg/Day | Lamotrigine 400 mg/Day | Lamotrigine 500 mg/Day
Number analyzed (Participants) | 149 | 67 | 49 | 46 | 164 | 84 | 34 | 18
percentage of participants | 70.5 | 59.7 | 20.4 | 13.0 | 80.5 | 67.9 | 38.2 | 16.7

17. Secondary Outcome: Change From Baseline to Week 56 in Hospital Anxiety and Depression Scale (HADS)
Description: Participant rated questionnaire with 2 subscales. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items; range: 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of symptoms. Scores relative to start of randomized treatment.
Time Frame: Baseline to Week 56
Population: FAS; N = number of participants with a HADS measurement at baseline and Week 56.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 237 | 238
scores on scale
  Anxiety | -0.3 (0.25) | -1.1 (0.25)
  Depression | -0.1 (0.23) | -0.7 (0.23)
Statistical Analysis 1: Comparison: Pregabalin vs Lamotrigine; Anxiety; model includes treatment and geographical cluster as fixed effects and respective baseline scores as a continuous covariate; Test type: Superiority or Other; p = 0.0025, ANCOVA; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [0.3 to 1.4]
Statistical Analysis 2: Comparison: Pregabalin vs Lamotrigine; Depression; model includes treatment and geographical cluster as fixed effects and respective baseline scores as a continuous covariate; Test type: Superiority or Other; p = 0.0186, ANCOVA; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [0.1 to 1.1]

18. Secondary Outcome: Medical Outcomes Study Sleep Scale (MOS-SS): Optimal Sleep Subscale
Description: MOS-SS: subject-rated instrument used to assess the key constructs of sleep over the past week; assesses sleep quantity and quality and is comprised 12 items yielding 7 subscale scores and 2 composite index scores. Optimal Sleep subscale is derived from sleep quantity average hours of sleep each night during the past week. Number of subjects with response Optimal if sleep quantity was 7 or 8 hours of sleep per night, and Non-optimal if average sleep was less than or greater than 7 to 8 hours per night. Analysis assesses the MOS-Sleep scale relative to the start of randomized treatment.
Time Frame: Week 8, Week 32, and Week 56
Population: FAS
Measure: Number; unit: participants
Arm/Group | Pregabalin | Lamotrigine
Number analyzed (Participants) | 330 | 330
participants
  Week 8: Optimal sleep | 195 | 173
  Week 8: Non-optimal sleep | 103 | 126
  Week 32: Optimal sleep | 167 | 155
  Week 32: Non-optimal sleep | 97 | 103
  Week 56: Optimal sleep | 152 | 145
  Week 56: Non-optimal sleep | 82 | 90
Statistical Analysis 1: Comparison: Pregabalin vs Lamotrigine; Week 8: dichotomized sleep assessment analyzed using a logistic regression model for repeated measures with fixed effects for treatment, geographical region, the average hours per night of sleep at baseline as a continuous covariate, time, and treatment-by-time interaction. The within subject covariance structure assumes an auto-regressive of order one covariance structure; Test type: Superiority or Other; p = 0.0683, Regression, Logistic; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.98 to 1.93]
Statistical Analysis 2: Comparison: Pregabalin vs Lamotrigine; Week 32: dichotomized sleep assessment analyzed using a logistic regression model for repeated measures with fixed effects for treatment, geographical region, the average hours per night of sleep at baseline as a continuous covariate, time, and treatment-by-time interaction. The within subject covariance structure assumes an auto-regressive of order one covariance structure; Test type: Superiority or Other; p = 0.5096, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.78 to 1.66]
Statistical Analysis 3: Comparison: Pregabalin vs Lamotrigine; Week 56 (termination): dichotomized sleep assessment analyzed using a logistic regression model for repeated measures with fixed effects for treatment, geographical region, the average hours per night of sleep at baseline as a continuous covariate, time, and treatment-by-time interaction. The within subject covariance structure assumes an auto-regressive of order one covariance structure; Test type: Superiority or Other; p = 0.6804, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.73 to 1.63]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin | Lamotrigine
Serious Adverse Events (participants affected / at risk) | 44/330 | 32/330
Other Adverse Events (participants affected / at risk) | 186/330 | 171/330
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=330) | Lamotrigine (N=330)
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Multiple endocrine adenomatosis Type II (Congenital, familial and genetic disorders) | 1 | 0
Parathyroid gland enlargement (Endocrine disorders) | 1 | 0
Entropion (Eye disorders) | 0 | 1
Trichiasis (Eye disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Chest pain (General disorders) | 0 | 1
Drowning (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Sudden unexplained death in epilepsy (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Vulvovaginitis (Infections and infestations) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 4
Foot fracture (Injury, poisoning and procedural complications) | 0 | 3
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 10 | 1
Dementia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Drug withdrawal convulsions (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 5 | 4
Grand mal convulsion (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 2 | 0
Partial seizures with secondary generalisation (Nervous system disorders) | 2 | 0
Postictal headache (Nervous system disorders) | 0 | 1
Spinal cord disorder (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 4 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Wernicke's encephalopathy (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Conversion disorder (Psychiatric disorders) | 1 | 1
Delirium tremens (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Vulval oedema (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1
Carpal tunnel decompression (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Ostectomy (Surgical and medical procedures) | 1 | 0
Splenectomy (Surgical and medical procedures) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=330) | Lamotrigine (N=330)
Vision blurred (Eye disorders) | 7 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 9
Abdominal pain upper (Gastrointestinal disorders) | 12 | 17
Constipation (Gastrointestinal disorders) | 9 | 5
Diarrhoea (Gastrointestinal disorders) | 12 | 13
Dyspepsia (Gastrointestinal disorders) | 8 | 12
Nausea (Gastrointestinal disorders) | 14 | 11
Toothache (Gastrointestinal disorders) | 9 | 4
Vomiting (Gastrointestinal disorders) | 7 | 8
Fatigue (General disorders) | 30 | 19
Pyrexia (General disorders) | 6 | 14
Influenza (Infections and infestations) | 14 | 12
Nasopharyngitis (Infections and infestations) | 15 | 21
Pharyngitis (Infections and infestations) | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 20 | 23
Weight increased (Investigations) | 22 | 7
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 6
Disturbance in attention (Nervous system disorders) | 7 | 6
Dizziness (Nervous system disorders) | 57 | 47
Headache (Nervous system disorders) | 75 | 73
Memory impairment (Nervous system disorders) | 8 | 13
Somnolence (Nervous system disorders) | 29 | 16
Anxiety (Psychiatric disorders) | 5 | 10
Depression (Psychiatric disorders) | 10 | 14
Insomnia (Psychiatric disorders) | 15 | 19
Sleep disorder (Psychiatric disorders) | 2 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 8
Rash (Skin and subcutaneous tissue disorders) | 12 | 18
Hypertension (Vascular disorders) | 4 | 7

LIMITATIONS AND CAVEATS:
Cox proportional hazards model for time to event (TTE) analyses; three summary statistics were not generated as median TTE will not exist if survival function (Kaplan-Meier product limit estimates) does not fall below 0.5 (post-hoc analysis).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.